CLINICAL TRIAL: NCT04480060
Title: Experience of an Emergency Intensive Care Unit During COVID-19 Pandemic: Retrospective Cohort Study
Brief Title: Experience of an Emergency Intensive Care Unit During COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ramazan Guven, Professor, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KSSEAH--EDCC
Record Dates: First submitted 2020-07-18; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: COVID-19 diagnostic PCR — Nasopharyngeal swab samples will be analyzed by PCR for COVID-19 DNA existence.

SUMMARY:
COVID-19, which emerged in China in December 2019, has become a pandemic with its spread to many countries of the world. Emergency departments also carried out an important part of the fight against pandemics in our country/Turkey. The emergency department including an intensive care unit is very few in this country/Turkey and the only hospital, which has an Emergency Intensive Care Unit (EICU) in Istanbul, is the study center. Therefore, this retrospective study aimed to provide useful information about how an effective EICU should be, especially how to use them during pandemic periods.

DETAILED DESCRIPTION:
COVID-19, which emerged in China in December 2019, has become a pandemic with its spread to many countries of the world. Emergency departments also carried out an important part of the fight against pandemics in our country/Turkey. The emergency department including an intensive care unit is very few in this country/Turkey and the only hospital, which has an Emergency Intensive Care Unit (EICU) in Istanbul, is the study center. Throughout the pandemic, many patients, including COVID-19 patients, were successfully followed up and discharged from EICU. With this study, the investigators expect to show the role of EICU during the pandemic. In addition, it will be seen that whether the patients, who are waiting for hospitalization or waiting for referral, are admitted to EICU faster and their treatments will be started promptly. Therefore, this retrospective study aimed to provide useful information about how an effective EICU should be, especially how to use them during pandemic periods.

ELIGIBILITY:
Inclusion Criteria:

* All patients who followed up in emergency department ICU with the diagnosis of COVID-19
* Accepted to participate with an informed consent

Exclusion Criteria:

* Patients under the age of 18 or more than 50 years
* declined to participate
* deaths caused by other than COVID-19

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients who followed up in emergency department ICU's of study centers with the diagnosis of COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
Mortality of the COVID-19 patients | 3 months
  Mortality of the COVID-19 patients who followed up by emergency department ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Seda Yilmaz Semerci, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No